

# **Clinical Investigation Plan for Medical Device Studies**

| | Digital care program for chronic shoulder |
|------------------------------|-------------------------------------------|
| F. II 444 6 | tendinopathy versus conventional physical |
| Full title of investigation: | therapy: a prospective, randomized |
| | controlled study |
| Version and date of Clinical | Version 1.4, 8 October 2020 |
| Investigation Plan (CIP): | version 1.4, 8 October 2020 |
| Sponsor: | SWORD Health |
| Sponsor CIP number: | SH-RCT-CS-US-01 |

# **REVISION HISTORY**

| Version | Date | Description | Author |
|---|---|---|---|
| 1.0 | 07/13/2020 | Original | FC and MM |
| 1.1 | 08/05/2020 | Content revision. Clarified procedures related to FC and MM participant intake and assessment. | |
| 1.2 | 08/26/2020 | Reviewed outcome measures and participant FC assessment procedures | |
| 1.3 | 09/22/2020 | Reviewed outcome measures, participant assessment procedures and clarified inclusion/Exclusion criteria | FC |
| 1.4 | 10/08/20202 | Reviewed exclusion criteria and conventional FC and SP PT treatment protocol | |

Version: 1.4

### **SIGNATURES**

The Principal Investigator (PI) and other personnel involved in the agree to perform the investigations and to abide by this CIP. The investigators agree to conduct the Investigation in compliance with all applicable laws and FDA Regulations Relating to Good Clinical Practice and Clinical Trials.

# Principal Investigator Sang (Sam) Pak, PT, DPT Assistant Professor, UCSF Signature Date: Sponsor Chief Medical Officer Fernando Correia, MD Chief Medical Officer, SWORD Health Technologies, Inc Signature Date: Sponsor Representative Virgílio Bento, PhD Chief Executive Officer, SWORD Health Technologies, Inc Signature


Date: 10/08/2020

Date:

### **SPONSOR**

# **Sponsor representative**

# **SWORD Health Technologies, Inc**

Virgílio Bento

1209 Orange Street

Wilmington, County of New Castle

Delaware 19801

Contact: +1 646-519-0638

Email: hello@swordhealth.com

# **STUDY INVESTIGATORS**

# **Principal Investigator**

# University of California San Francisco

Sam Pak

Box 0736

San Francisco

California 94158

Contact: +1 646-519-0638 Email: sam.pak@ucsf.edu


# TABLE OF CONTENTS

| REV | ISION HISTORY | II |
|-------|--------------------------------------------------|-----|
| SIGN | NATURES | III |
| SPO | NSOR | IV |
| STUI | DY INVESTIGATORS | IV |
| 1. | BACKGROUND | 1 |
| 1. | SWORD HEALTH DIGITAL CARE PROGRAMS | 3 |
| 2. | SYSTEM TECHNICAL SPECIFICATIONS | 4 |
| 3. | SECURITY AND DATA STORAGE | 5 |
| 3.1 | DATABASE | 5 |
| 3.2 | WEB PORTAL | 5 |
| 3.3 | WEBSITE | 5 |
| 3.4 | MOBILE APP | 6 |
| 4. | STUDY OBJECTIVE | 6 |
| 5. | STUDY HYPOTHESIS | 6 |
| 6. | STUDY DESIGN | 6 |
| 7. | STUDY OUTCOMES | 6 |
| 8. | SAMPLE SIZE ESTIMATION | 8 |
| 9. | INCLUSION/EXCLUSION CRITERIA | 8 |
| 9.1. | INCLUSION CRITERIA | 8 |
| 9.2. | EXCLUSION CRITERIA | 9 |
| 10. | CANDIDATE IDENTIFICATION AND PROCEEDINGS | 9 |
| 11. | PROCESS OF CONSENT | 10 |
| 12. | ALLOCATION & BLINDING | 10 |
| 13. | INTERVENTION | 11 |
| 13.1. | DIGITAL PROGRAM | 11 |
| 13.2. | CONVENTIONAL PT | 12 |
| 14. | ASSESSMENTS | 12 |
| 15. | STATISTICAL ANALYSIS PLAN | 16 |
| 16. | RISKS AND BENEFITS | 16 |
| 17. | CONFIDENTIALITY | 17 |
| 18. | REFERENCES | 18 |
| ANN | EX 1 - INFORMED CONSENT FORM | 24 |
| ANN | EX 2- DIGITAL THERAPEUTIC EXERCISE PROTOCOL | 6 |
| ANN | EX 3- CONVENTIONAL THERAPEUTIC EXERCISE PROTOCOL | 14 |

### 1. BACKGROUND

Shoulder pain is highly prevalent, being the third main complaint in primary care settings. <sup>1–3</sup> There is a wide range of reported incidence and prevalence rates, with a median of 24.8% of adults reporting shoulder pain every month.<sup>4</sup> In developed countries, 1% of adults annually consult a primary care provider due to shoulder pain.<sup>2,5</sup>

Around 65 to 70% of shoulder pain complaints involve problems in the rotator cuff (RTC) tendons, 1,6 with incidence rising higher after the 4th decade of life. 1,7-9 Abundant data from across the world is available on the prevalence of RTC pathologies. 6,10-16

RTC dysfunction represent a huge burden for healthcare systems, insurance companies and employers alike.<sup>1,17</sup> Shoulder problems account for 2.4% of all general practitioner consultations in the UK. 18 and 4.5 million visits to physicians annually in the USA. 19 One study in the UK<sup>20</sup> estimated that nearly £310 million is spent on medical appointments in the first 6 months of shoulder pain onset, and additional costs of surgical procedures are estimated at approximately £30 million/year, with up to 50% of these costs related to sick leave from paid employment. More than 300,000 surgical repairs for RTC pathologies are performed annually in the USA, and the annual financial burden of RTC management was also estimated at \$3 billion.<sup>21</sup>

A myriad of international clinical practice guidelines have been put forth over the years, outlining the management of pain-causing shoulder disorders. 22-26 Most causes of mild-to-moderate and gradual onset shoulder pain are treated initially with conservative care. Indeed, many recent studies and systematic reviews, as well as the American Academy of Orthopaedic Surgeons guidelines, support that firstly the patient should be directed to a physical therapy (PT) program and not surgery. <sup>26–30</sup> For some specific conditions (e.g., symptomatic small to medium full-thickness RTC tears), strong evidence further supports that both PT and operative treatment attain significant improvements in patient-reported outcomes.<sup>26</sup> Of note, another systematic review on treatment options for shoulder pain suggests that passive modalities, such as manual therapy, electrotherapy and taping should be avoided as mono-therapy but that they could, in specific cases, provide

Date: 10/08/2020

Version: 1.4 1 additional benefit when utilized in conjunction with therapeutic exercise programs.<sup>31</sup> This suggests that the exercise component of PT is fundamental in the treatment of painful shoulder disorders.

Regarding rehabilitation setting, some studies show that home-based therapy, based on exercise, could be as effective as conventional PT interventions. 32,33 This is in line with the recent trends in healthcare delivery, moving away from inpatient care and towards home-based care with the intent of improving costeffectiveness. Furthermore, the need for home-based digital solutions is now felt more acutely than ever, in the face of the current pandemic. <sup>34–36</sup> In this context, solutions enabling home-based rehabilitation without requiring real-time human supervision can be key to improving effectiveness and lowering costs, while keeping all stakeholders safe. Indeed, there are studies demonstrating the potential<sup>37–39</sup> and costeffectiveness<sup>40</sup> of shoulder postoperative care and rehabilitation through telehealth solutions.

However, while evidence is growing that digital therapeutics (DTx) can improve outcomes, personalize care and decrease costs, 41 there is still much ground to be explored in the field of digital therapy following RCR. 42,43 Several studies can be found on the validation/development of systems/algorithms for monitoring shoulder motion to assist clinicians on patient evaluation 44,45 but these do not meet the aforementioned needs and cannot be considered digital therapeutics.

There have been some advances on new technologies for shoulder rehabilitation, namely using wearable sensors<sup>43</sup> and augmented reality.<sup>46</sup> Of note, some of these studies focus on systems based on inertial motion trackers that can be used by the patient at home, under remote monitoring from the physical therapist. However, these are either in very preliminary stages of development or validation, <sup>47–51</sup> with no clinical validation studies performed, or are directed at rehabilitation after stroke. 43,46

SWORD Health has developed a novel motion tracking-based digital biofeedback system for home-based physical rehabilitation - SWORD Phoenix®- which is an FDA-listed class II medical device. The company has previously conducted two pilot studies (NCT03047252; NCT03045549) comparing a digital therapy program using this device against conventional face-to-face physical therapy. These studies have proven the feasibility, safety and effectiveness of this digital therapeutic on rehabilitation after total knee and hip arthroplasty. 52-54

This is a single-center, prospective, randomised, controlled study, with two parallel groups, designed to assess the clinical impact of a digital exercise program against conventional rehabilitation for shoulder tendonitis. The hypothesis is that all the clinical outcomes measured

will significantly improve after the program, and patients using this novel system will attain at

least the same outcomes than the ones attained by the conventional PT group.

2. SWORD HEALTH DIGITAL CARE PROGRAMS

SWORD Health's Digital Care programs address the three pillars of musculoskeletal care:

therapeutic exercise, patient education and cognitive behavioural therapy (CBT).

The exercise component is delivered through a digital feedback system - SWORD Phoenix®-

which is an FDA-listed class II medical device. This device uses motion tracking technology to

digitize motion and provide real-time biofeedback on performance during exercise execution (see

more below). This allows individuals to perform independent exercise sessions at home without

the need for constant face-to-face therapist supervision, while still being remotely monitored

(asynchronously) through a cloud-based Portal.

The safety and effectiveness of digital exercise programs performed with this device, in a home-

based scenario, have already been demonstrated for recovery after total knee and hip

arthroplasty. 53–55 In these studies, where digital programs based on this device were compared with

conventional PT, the clinical outcomes were superior in the digital group. These results were

explained by (a) the positive impact of a kinematic biofeedback tool on patient performance,

especially regarding error correction and stimulation of a greater range of motion; (b) patient

empowerment regarding their rehabilitation process; (c) high patient engagement through the use

of gamification strategies; (d) the positive effect of remote monitoring on patient effort and (e) the

availability of objective data for clinical review, enabling data-driven decisions.

The education component is delivered through a smartphone app. Through this app, each

individual is presented with educational content on their condition, in the form of small articles

curated by SWORD's clinical team, focusing on subjects ranging from anatomy and physiology,

pain, exercise and fear avoidant behaviours.

The CBT component takes the form of an 8-week program based on third-generation CBT

techniques, particularly Mindfulness Based Stress Reduction, Acceptance and Commitment

Date: 10/08/2020

Version: 1.4 3

Therapy and Compassion-based therapy. The program is presented to individuals through email,

with links to short, pre-recorded, self-guided, meditation sessions, as well as written mindfulness

exercises called "habit releasers".

3. SYSTEM TECHNICAL SPECIFICATIONS

**SWORD Phoenix**® is a proprietary, 510(K) exempt, class I medical device, with CE mark, which

is composed of the following three interconnected components:

■ Motion trackers, placed on body segments using Velcro® straps. Each motion tracker is placed in a

specific position. To assist in the correct placement of the motion trackers, both the trackers and the

matching straps are color-coded. The motion trackers' setup varies according to each therapy.

Mobile App, that comes pre-installed on a tablet, that guides the patient in each exercise session. Before

each exercise, the patient is presented with a real-life video and audio explanation of that exercise. The

execution interface is subsequently shown. This screen features: a) a progress bar; b) a repetition

counter; c) a star counter and d) a timer displaying time left in the exercise. A correct repetition is

defined as a movement starting at the baseline and reaching or surpassing the specified target, without

violating movement or posture constraints. In case the patient violates a constraint, a message is

prompted showing which movement error was performed, so that the patient can correct the movement

in the following attempts. For each correct repetition, the patient earns from 1 to 5 stars, depending on

the range of motion of that specific movement in comparison to normative values for that movement.

At the end of each session, the patient is presented with a summary of the number of completed

repetitions and stars, as well as with badges rewarding him for the progresses achieved in each exercise.

• Web-based Portal that allows the clinical team to generate new patient profiles and create exercise

sessions for each patient. To prescribe a session, the clinician needs to select the exercises, number of

sets and number of repetitions. When a patient performs a session, the results are uploaded to the

platform and available for review. Based on this information, the clinical team can edit the parameters

of each exercise according to patient performance and progress.


Date: 10/08/2020

4

4. SECURITY AND DATA STORAGE

4.1 DATABASE

The networks where SWORD Health's infrastructure is hosted are maintained by Google and are

included in Google Cloud Platform's SOC2 and HITRUST certifications. Security-related

configurations are registered and verified periodically.

Collected data is stored in databases that are only accessible to SWORD's Application

Programming Interface (API), and Personal Health Information (PHI) is individually encrypted

inside this database. Separate databases are used for development, OA, and production

environments.

4.2 WEB PORTAL

Data is secured in transit to SWORD's Application Programming Interface (APIs) due to enforced

application of TLS 1.2 or above. Additionally, a web application firewall protects our servers from

Cross-site Scripting (XSS) and SQL Injection attacks.

Access to SWORD's Web Portal is provided only to individuals who have a valid work contract

with SWORD Health and have a role within the company that allows them to use the platform (i.e.

PTs and IT support).

Access control mechanisms ensure that only authorized users have access to PHI and different

functions are mapped to different roles within the platform (i.e. IT support personnel only have

access to de-identified data).

4.3 WEBSITE

SWORD's Onboarding Website does not have a login function as it works only as a registry

platform and user accounts are created in SWORD's Web Portal. Data is secured in transit to

SWORD's Application Programming Interface (APIs) due to enforced application of TLS 1.2 or

above. Additionally, a web application firewall protects our servers from Cross-site Scripting

(XSS) and SOL Injection attacks.


5

4.4 MOBILE APP

For an individual to access the mobile app in the medical device, their profile must be created in

SWORD's Web Portal. Upon profile creation, the individual is attributed a unique QR card that is

shipped together with the medical device kit. Upon the first usage, the individual is required to set

a personal pin code (two-factor authentication is employed, as the user must scan their QR code

and input a confirmation code sent by text message. This is required for the first login, with

subsequent logins being done by presenting the pin and the QR card. Each session expires within

24 hours, requiring the individual to present these again if >24 hours have passed since the last

usage.

Transport Layer Security (TLS) protocols are applied on every connection to ensure secure data

transmission between the mobile app and the Database. Additionally, data stored in the device is

also encrypted.

5. STUDY OBJECTIVE

To assess the clinical outcomes of a digital program for chronic shoulder tendonitis versus

conventional. PT.

6. STUDY HYPOTHESIS

The digital program will be associated with at least the same outcomes as conventional PT.

7. STUDY DESIGN

Prospective, single-center, parallel-group, randomised controlled study.

8. STUDY OUTCOMES

**8.1 Primary Outcome** 

Impact on physical function and symptoms measured through the shortened Disabilities of the

Arm, Shoulder and Hand questionnaire (QuickDASH) between baseline and 8 weeks.


6

8.2 Secondary Outcomes

The secondary outcomes will include the following:

a) Impact on shoulder range of motion

Shoulder range of motion will be measured in the following exercises: shoulder flexion; shoulder

abduction and external shoulder rotation at 90 degrees of abduction.

b) Impact on Pain

Measured through the following question: "On a scale of 0 to 10, where 0 is no pain and 10 the

worst pain imaginable, how would you rate your pain in the last 24 hours?"

c) Interest in undergoing surgery

Measured through the following question: "On a scale of 0 to 10, where 0 is not at all and 10 is

extremely interested, how interested are you in undergoing shoulder surgery in the next 12

months"?

d) Medication consumption

Measured through the following questions:

i. "Are you taking any medication for your shoulder pain?";

ii. "If yes, on how many days in a week, on average, are you taking medication for your shoulder

pain"

e) Impact on fear avoidance beliefs

Measured by: Patient-reported questionnaire (Fear Avoidance Beliefs Questionnaire- FABQ)

f) Impact on anxiety and depression

Measured by the General Anxiety Disorder-7 scale and Patient Health Questionnaire-9 scale

g) Impact on work productivity and activity impairment

Measured through Work Productivity and Activity Impairment Questionnaire: Specific Health

Problem v2.0 (WPAI:SHP)


Date: 10/08/2020

7

h) Satisfaction with social roles and discretional social activities

Measured through the Patient Reported Outcomes Measurement Information System

Computerized Adaptive Test (PROMIS-CAT) scales: Ability to participate in social roles and

activities (version 2.0) and satisfaction with social roles and activities (version 2.0).

i) Patient engagement

Measured through: g.1) adherence to exercise sessions; g.2) drop-out rates; g.3) treatment

intensity (i.e. total number of exercise minutes)

j) Patient satisfaction

Measured through the Net Promoter Score, by asking participants the following question: "On a scale

from 0 to 10, how likely are you to recommend this program to a friend or colleague?"

9. SAMPLE SIZE ESTIMATION

Sample size estimation calculations were performed taking into consideration the primary outcome

measure – the QuickDASH. In a sample of 57 patients with shoulder tendon disorders treated with

SWORD Health's medical device in the context of work-related conditions, the mean and standard

deviation of the QuickDASH scale at baseline was of 59 and 19 points respectively. A Minimal

Detectable Difference (MDD) of 11.2 points was considered, based on the psychometric properties

of the scale.<sup>56</sup> Considering a power of 80%, a two-sided 0.05 significance level and a 10% dropout

rate, 80 (40+40) patients would be necessary to detect a 11.2 points difference between the two

groups.

10. INCLUSION/EXCLUSION CRITERIA

a. Inclusion Criteria

a) Subjects aged between 18 and 80 years of age at enrolment

b) Reporting intermittent or persistent shoulder pain for at least 6 weeks, and/or present at least

50% of the time in the past 6 months

c) Lack of visual/audio or cognitive impairment interfering with the ability to understand or

comply with the program


8

### b. Exclusion Criteria

- a) Non-English speaking
- b) Residing outside greater SF area
- c) Known pregnancy
- d) Submitted to spinal surgery less than 3 months ago
- e) Symptoms and/or signs indicative of possible infectious disorder
- f) Referred pain from spine and/or thoracic outlet syndrome
- g) Active cancer diagnosis or undergoing treatment for cancer
- h) Cardiac, respiratory or other known disorder incompatible with at least 20 minutes of light to moderate physical activity
- i) Concomitant neurological disorder (e.g. stroke, multiple sclerosis, Parkinson's disease)
- j) Dementia or psychiatric disorders precluding patient from complying with a home-based exercise program
- k) Illiteracy and/or serious visual or auditory impairment interfering with communication or compliance

Additionally, any patient undergoing a PT program for shoulder pain will be required to stop ongoing programs to enroll in the study.

### 11. CANDIDATE IDENTIFICATION AND PROCEEDINGS

Patient recruitment will primarily be done through the use of UCSF electronic health record (EHR) recruitment services from the Clinical and Translational Service Institute (CTSI) to assist with targeting and identification of potentially eligible participants. As an "honest broker" of the EHR data, the service is designed to protect patient privacy and offer more efficient way to recruit eligible participants that meets the study's inclusion/exclusion criteria. The cohort of patients scheduled to receive physical therapy services will be identified and pre-screened by CTSI to ensure potential participants are eligible to meet the initial study's criteria. Once patients have been identified, they are flagged from their appointments for physical therapy services at the UCSF Outpatient Patient Faculty, and will be evaluated in-person as part of their regular initial scheduled visit (i.e. evaluation visit). At the time of this visit, potential participants will be assessed by one of the co-investigators to also ensure that participants meet the cognitive and mental capacity

requirements. Once the criteria are met, investigator will present the study and invite the patient to

participate and provide consent. The participant's screening survey data will be collected and be

randomized to one of the two arms, coordinated by the study coordinator. All study-related

information will be stored by electronic data capturing (EDC) system.

To centralize all study-related information, a commercially available electronic data capturing

(EDC) system will be used.

Following the identification of a potential candidate, the investigator will enter the EDC portal and

fill the screening survey. If the patient is eligible (i.e. meets inclusion criteria and does not have

any exclusion criteria) the investigator will present the study and invite the patient to participate

and provide consent.

12. PROCESS OF CONSENT

The study will be presented verbally to potential participants by a study investigator, in a face-to-

face meeting. Adequate time will be allowed for the candidate to clarify any doubts about the

study, following which the eConsent form will be sent through the EDC platform to the participant

and investigator, for signature. The study consent form (Annex 1) will then be signed by the

participant and the investigator collecting consent, and stored in the EDC platform.

13. ALLOCATION & BLINDING

Patients will be randomly allocated to one of two groups, using random permuted blocks of 6.

After eConsent collection, the investigator will enter the EDC portal and proceed with

randomisation (also built into the EDC). Following randomisation, the investigator will contact

the person responsible for the rehabilitation program in each group to allocate the participant to

the respective study arm. Blinding of investigators and patients regarding allocation arm will not

be possible, given the nature of the intervention. Analysis of study results will be performed by an

independent statistician at UCSF.


Date: 10/08/2020

10

### 14. Intervention

### a. Digital program

Patients in the digital intervention group will benefit from an 8-week program composed of therapeutic exercise, education and cognitive behavioural therapy (CBT) program provided by SWORD Health. These patients will be referred to SWORD Health by the investigator who identified the candidate. SWORD Health will then assign a physical therapist to each patient. The physical therapist will contact the patient for onboarding and will manage the case.

Patients in this group will performed home-based rehabilitation sessions using SWORD Phoenix<sup>®</sup>, under remote monitoring by a physical therapist. Participants will be provided with a tablet computer with a SWORD mobile app installed, along with two inertial motion trackers (each comprised of a gyroscope, an accelerometer and a magnetometer) to be placed on chest, upper arm and wrist, respectively. These trackers enable precise movement quantification, feeding the mobile app, which guides the patient through the session, providing video and audio instructions before each exercise, as well as real-time audio and video biofeedback during the exercise. On the other end, the clinical teams are allowed to remotely monitor results and prescribe/edit exercise sessions through a web-based portal.

The exercise component will follow the protocol outlined in **Annex 2**, which can however be adapted by the physical therapist to the specific needs of the participant. Participants will be asked to start with three 20 min sessions per week, building gradually to three 30 min sessions per week. Participants will not be excluded from the study in case of lower adherence, but will not be included in the per-protocol analysis if they perform less than 21 sessions over the course of 8 weeks.

Participants in this group will be considered as dropouts if they: a) choose to abandon the study; b) do not engage in any exercise session for at least fourteen consecutive days.

The educational component will be delivered automatically through a smartphone app (available for iOS and Android), and will take the form of small educational texts that will be released


periodically to the participant. This component is not mandatory per protocol, but metrics on user

engagement will be measured.

The CBT program will take the form of a self-paced program consisting of written and pre-

recorded audio materials. An email will be sent weekly by the physical therapist to the participant,

during the 8 weeks of the program. Each email will contain an introductory text describing the

objectives for that week, as well as a link to that week's audio session and a PDF attachment with

self-guided exercises. The CBT component is not mandatory per protocol, but metrics on user

engagement will be measured.

b. Conventional PT

Patients in this group will benefit from a 8-week program consisting of two 30 min face-to-face

PT sessions per week in an outpatient clinic setting, for a total of 16 sessions. The program will

follow the principles outlined in Annex 3, which includes commonly used interventions adapted

by the physical therapist to the specific needs of the participant.

Participants in this group will be excluded from the per protocol analysis if they complete less than

14 sessions over 8 weeks. Participants in this group will be considered as dropouts if they: a)

choose to abandon the study; b) miss four consecutive scheduled PT sessions.

In addition to the face-to-face sessions, PTs will also be communicating with participants in this

group through a secure messaging system (Mychart) used at UCSF or, alternatively, through a

telephone check-ins (10-15 min calls, up to twice per week).

15. PARTICIPANT ASSESSMENTS

Patients will be assessed at baseline, 4 and 8 weeks.

**Baseline Assessment** 


12

This assessment will involve a face-to-face visit, where the following information will be collected:

- a) date of birth
- b) gender
- c) height & weight
- d) body mass index
- e) formal education (years of schooling)
- f) job type
- g) previous shoulder surgery (> 3 months ago)
- h) Working status
- i) Geocodes/zip
- i) Race/ethnicity
- k) Age

The following outcomes will also be assessed in this visit: a) Shoulder Range of Motion; b) PROMIS CAT measures.

Shoulder Range of Motion will be measured in the following movements: 1) shoulder flexion; 2) shoulder abduction; 3) external rotations with shoulder abducted at 90 degrees. The participant will be asked to perform three non-painful repetitions of each movement, in a standing position. The investigator will measure the maximum joint angle attained by the participant, using a digital goniometer in each repetitions. The highest of the three values will be considered.

Regarding satisfaction with social role and ability to participate in social roles and activities, these will be collected through PROMIS CAT v2.0. These will be collected onsite, and the results will then be transferred by the investigator to the eCRF.

Assessment of primary outcome, as well as the remaining secondary outcomes will be performed through an electronic questionnaire to be filled by participants, through the EDC system. These will need to be filled within 5 consecutive days, counting from the date they are sent to the participant. To promote compliance with this schedule, whenever the deadline is approaching, automatic email reminders will be sent to participants. Participants will be excluded from the study

for protocol breach in case they don't fill in the assessment forms. Upon completion of the baseline

form, participants in the study will receive a stipend of \$25.

Additional measurements of upper limb function and tri-dimensional motion will also be

performed at the onsite visit by the clinician, using a motion capture system. These will not be

considered in the outcomes of this study, but will be made available for post-hoc analysis.

**Interim assessment (4 weeks)** 

Participants will be required to complete a questionnaire similar to the baseline assessment, within

a 5-day window beginning at the start of week 4. These assessments will include all the information

pertaining to the primary and secondary outcomes, except for those that are collected through a

face-to-face assessment. These (shoulder range of motion and PROMIS CAT measures) will not

be collected on this assessment. Upon completion of this form, participants in the study will receive

a stipend of \$25.

Final assessment (8 weeks)

This assessment will involve a face-to-face visit, where the following outcomes will be assesed:

a) shoulder Range of Motion; b) PROMIS CAT measures and c) Participant satisfaction (Net

Promoter Score). Shoulder Range of Motion and PROMIS CAT measures will be assessed using

a similar methodology to the one descried for the baseline assessment.

Participants will also be required to complete a questionnaire similar to the baseline and interim

assessments, within a 5-day window beginning at the start of week 4. These assessments will

include all the information pertaining to the primary and secondary outcomes, except for those that

are collected in the face-to-face visit. Upon completion of this form, participants in the study will

receive a stipend of \$25.


Date: 10/08/2020

14

Additional measurements of upper limb function and tri-dimensional motion will also be

performed at the onsite visit by the clinician, using a motion capture system. These will not be

considered in the outcomes of this study, but will be made available for post-hoc analysis.

**Engagement assessment** 

For participants on the digital group, engagement and usage metrics of the educational and CBT

components will also be collected automatically.

Additionally, the following activity log will be collected from patient's Electronic medical records

and time stamps, as well as paper survey (or, in the case of the digital group, sent to the study

coordinator via email, with the participant identified only by the study ID), to be entered into EDC

portal by study coordinator:

1. Face-to-face visits registry (dates, times and duration)

2. Remote sessions registry (dates, times and duration)

3. Number and duration of contacts between PT and participant (emails, text messages, phone and

videocalls)

4. Total time spent on remote monitoring of the patient (digital group only)

Adverse events

In any event during the course of the study if subjects experience adverse effects of both internal

(on-site) and external (off-site) events, a prompt reporting to the UCSF Human Research

Protection Program (HRPP)/institutional review board (IRB) and to the sponsor of the study will

take place. This includes any unanticipated problems involving risk to subjects noted in the study.

The safety plan in IRB will contain protocol to help with communication and procedures that are

in place to monitor and report adverse events should they occur. The investigators will accurately

document causality assessment to their best knowledge and follow-up of all definite, probable, or

unrelated adverse events to the study and safety-related information.

**Care continuity** 

To ensure that quality of care is not compromised throughout the study, all subjects from both

Version: 1.4 15 Date: 10/08/2020

groups will be assessed at the final appointment to determine whether further care is warranted. If

subjects require additional physical therapy services or follow-up back to the physician, the

primary investigator will coordinate with UCSF physical therapist to ensure continuity of care or

proper closure of their care are complete.

16. STATISTICAL ANALYSIS PLAN

To assess differences in clinical and demographic variables of the patients allocated to the two

study groups, independent samples t test or Mann-Whitney U test will be used for quantitative

variables. For categorical variables, Chi-square test or Fisher's exact test will be used.

Outcome analysis will be performed using both an intention to treat analysis and a per-protocol

analysis.

The overall impact of the intervention on the primary and secondary outcomes will be assessed

considering both the results at the 8-week assessment as well as change from baseline.

Differences between interventions will be evaluated using independent samples t test or Mann-

Whitney U test. For non-normally distributed variables, the magnitude of the difference in the

medians will be assessed using Hodges-Lehman estimator. Additionally, a repeated measures

ANOVA will also be performed, with group as an independent factor and time as a within-subjects

factor. When necessary, logarithmic transformation will be performed to obtain normally

distributed variables. In all analysis, a significant level of 0.05 will be considered.

17. RISKS AND BENEFITS

Participants in this clinical study will be allocated to one of two treatment groups. In any case, they

will be receiving an evidence-based treatment program tailored to their condition, overseen by

physicians and physical therapists. Participants in the digital care program will be performing the

exercise component using a certified medical device for its intended purpose. Therefore,

participants are not running additional risks by participating in this study.

Exercise programs can, however, be associated with temporary pain or discomfort as expected

from the typical treatment. In the digital care group, pain and fatigue scores will be asked at the

end of each session, and this information is relayed to the physical therapist assigned to the

Date: 10/08/2020


participant, who will contact the patient in case of excessive pain or fatigue. In the conventional

PT group, sessions will be performed under direct supervision from a physical therapist. In any

case, both participants and physical therapists will be instructed to contact the study investigators

in case of an adverse event.

As to the benefits, by participating in this study, participants may experience reduction in pain,

improvement in function, mood and general well-being. However, the effects may vary from

person to person, and therefore substantial improvements cannot be guaranteed.

18. CONFIDENTIALITY

PHI will be shared with individuals and organizations that conduct or watch over this research,

including:

- The research sponsor

- People who work with the research sponsor

- Government agencies, such as the Food and Drug Administration

- The Institutional Review Board (IRB) that reviewed this research

Data used for dissemination of study results will be de-identified before publication.


17

### 19. REFERENCES

- 1. Edwards P, Ebert J, Joss B, Bhabra G, Ackland T, Wang A. Exercise Rehabilitation in the Non-Operative Management of Rotator Cuff Tears: a Review of the Literature. *Int J Sports Phys Ther*. 2016;11(2):279-301.
- 2. Mitchell C, Adebajo A, Hay E, Carr A. Shoulder pain: Diagnosis and management in primary care. *Bmj.* 2005;8(November):331-1124. doi:10.1007/BF00320147
- 3. Lewis JS. Rotator cuff tendinopathy/subacromial impingement syndrome: Is it time for a new method of assessment? *Br J Sports Med.* 2009;43(4):259-264. doi:10.1136/bjsm.2008.052183
- 4. Luime JJ, Koes BW, Hendriksen IJM, et al. Prevalence and incidence of shoulder pain in the general population; a systematic review. *Scand J Rheumatol*. 2004. doi:10.1080/03009740310004667
- 5. Tekavec E, Jöud A, Rittner R, et al. Population-based consultation patterns in patients with shoulder pain diagnoses. *BMC Musculoskelet Disord*. 2012. doi:10.1186/1471-2474-13-238
- 6. Thomson S, Jukes C, Lewis J. Rehabilitation following surgical repair of the rotator cuff: a systematic review. *Physiotherapy*. 2016;102(1):20-28. doi:10.1016/j.physio.2015.08.003
- 7. Hawkins RJ, Morin WD, Bonutti PM. Surgical treatment of full-thickness rotator cuff tears in patients 40 years of age or younger. *J Shoulder Elbow Surg*. 1999;8(3):259-265.
- 8. Mall NA, Lee AS, Chahal J, et al. An evidenced-based examination of the epidemiology and outcomes of traumatic rotator cuff tears. *Arthrosc J Arthrosc Relat Surg*. 2013. doi:10.1016/j.arthro.2012.06.024
- 9. Tempelhof S, Rupp S, Seil R. Age-related prevalence of rotator cuff tears in asymptomatic shoulders. *J Shoulder Elb Surg*. 1999;8(4):296-299. doi:10.1016/S1058-2746(99)90148-9
- 10. Sambandam SN, Khanna V, Gul A, Mounasamy V. Rotator cuff tears: An evidence based approach. *World J Orthop*. 2015. doi:10.5312/wjo.v6.i11.902
- 11. Grant HJ, Arthur A, Pichora DR. Evaluation of interventions for rotator cuff pathology: A systematic review. *J Hand Ther*. 2004. doi:10.1197/j.jht.2004.02.013
- 12. Littlewood C, May S, Walters S. Epidemiology of Rotator Cuff Tendinopathy: A Systematic Review. *Shoulder Elb.* 2013. doi:10.1111/sae.12028


- 13. Bey MJ, Song HK, Wehrli FW, Soslowsky LJ. Intratendinous strain fields of the intact supraspinatus tendon: The effect of glenohumeral joint position and tendon region. *J Orthop Res.* 2002;20(4):869-874. doi:10.1016/S0736-0266(01)00177-2
- 14. Littlewood C, Bateman M. Rehabilitation following rotator cuff repair: a survey of current UK practice. *Shoulder Elb.* 2015;7(3):193-204. doi:10.1177/1758573215571679
- 15. Ross D, Maerz T, Lynch J, Norris S, Baker K, Anderson K. Rehabilitation following arthroscopic rotator cuff repair: A review of current literature. *J Am Acad Orthop Surg*. 2014. doi:10.5435/JAAOS-22-01-1
- 16. Factor D, Dale B. Current concepts of rotator cuff tendinopathy. *Int J Sports Phys Ther*. 2014;9(2):274-288.
- 17. Mather III RC, Koenig L, Acevedo D, et al. The Societal and Economic Value of Rotator Cuff Repair. *J Bone Jt Surg.* 2013;95:1993-2000.
- 18. Linsell L, Dawson J, Zondervan K, et al. Prevalence and incidence of adults consulting for shoulder conditions in UK primary care; patterns of diagnosis and referral. *Rheumatology*. 2006. doi:10.1093/rheumatology/kei139
- 19. Oh LS, Wolf BR, Hall MP, Levy BA, Marx RG. Indications for Rotator Cuff Repair. *Clin Orthop Relat Res.* 2007. doi:10.1097/blo.0b013e31802fc175
- 20. Littlewood C, May S. A contractile dysfunction of the shoulder. *Man Ther*. 2007. doi:10.1016/j.math.2005.11.002
- 21. Aurora A, McCarron J, Iannotti JP, Derwin K. Commercially available extracellular matrix materials for rotator cuff repairs: State of the art and future trends. *J Shoulder Elb Surg.* 2007. doi:10.1016/j.jse.2007.03.008
- New Zealand Guidelines Group. The Diagnosis and Management of Soft Tissue Shoulder Injuries and Related Disorders: Best practice Evidence-Based Guidelines. *Accid Compens Corp.* 2004.
- 23. Hanchard NCA, Goodchild L, Thompson J, O'Brien T, Davison D, Richardson C. Evidence-based clinical guidelines for the diagnosis, assessment and physiotherapy management of contracted (frozen) shoulder: Quick reference summary. *Physiotherapy*. 2012. doi:10.1016/j.physio.2012.01.001
- 24. Kelley MJ, Shaffer MA, Kuhn JE, et al. Shoulder Pain and Mobility Deficits: Adhesive Capsulitis. *J Orthop Sport Phys Ther*. 2013. doi:10.2519/jospt.2013.0302


- 25. Oliva F, Piccirilli E, Bossa M, et al. I.S.Mu.L.T Rotator cuff tears guidelines. *Muscles Ligaments Tendons J.* 2015. doi:10.11138/mltj/2015.5.4.227
- 26. American Academy of Orthopaedic Surgeons. Management of Rotator Cuff Injuries Clinical Practice Guideline. 2019.
- 27. Beaudreuil J, Dhénain M, Coudane H, Mlika-Cabanne N. Clinical practice guidelines for the surgical management of rotator cuff tears in adults. *Orthop Traumatol Surg Res.* 2010. doi:10.1016/j.otsr.2010.02.002
- 28. Gebremariam L, Hay EM, Koes BW, Huisstede BM. Effectiveness of surgical and postsurgical interventions for the subacromial impingement syndrome: A systematic review. *Arch Phys Med Rehabil*. 2011. doi:10.1016/j.apmr.2011.06.006
- 29. Pedowitz RA, Yamaguchi K, Ahmad CS, et al. Optimizing the management of rotator cuff problems. *J Am Acad Orthop Surg*. 2011. doi:10.5435/00124635-201106000-00007
- 30. Seida JC, LeBlanc C, Schouten JR, et al. Systematic review: Nonoperative and operative treatments for rotator cuff tears. *Ann Intern Med.* 2010. doi:10.7326/0003-4819-153-4-201008170-00263
- 31. Yu H, Cote P, Shearer HM, et al. Effectiveness of Passive Physical Modalities for Shoulder Pain: Systematic Review by the Ontario Protocol for Traffic Injury Management Collaboration. *Phys Ther*. 2015. doi:10.2522/ptj.20140361
- 32. Walther M, Werner A, Stahlschmidt T, Woelfel R, Gohlke F. The subacromial impingement syndrome of the shoulder treated by conventional physiotherapy, self-training, and a shoulder brace: Results of a prospective, randomized study. *J Shoulder Elb Surg.* 2004. doi:10.1016/j.jse.2004.02.002
- 33. Kuhn JE. Exercise in the treatment of rotator cuff impingement: A systematic review and a synthesized evidence-based rehabilitation protocol. *J Shoulder Elb Surg*. 2009. doi:10.1016/j.jse.2008.06.004
- 34. Eccleston C, Blyth FM, Dear BF, et al. Managing patients with chronic pain during the COVID-19 outbreak: considerations for the rapid introduction of remotely supported (eHealth) pain management services. *Pain*. 2020. doi:10.1097/j.pain.000000000001885
- 35. Parisien RL, Shin M, Constant M, et al. Telehealth Utilization in Response to the Novel Coronavirus (COVID-19) Pandemic in Orthopaedic Surgery. *J Am Acad Orthop Surg*. 2020. doi:10.5435/JAAOS-D-20-00339


- 36. Wosik J, Fudim M, Cameron B, et al. Telehealth transformation: COVID-19 and the rise of virtual care. *J Am Med Informatics Assoc*. 2020. doi:10.1093/jamia/ocaa067
- 37. Kane LT, Thakar O, Jamgochian G, et al. The role of telehealth as a platform for postoperative visits following rotator cuff repair: a prospective, randomized controlled trial. *J Shoulder Elb Surg.* 2020. doi:10.1016/j.jse.2019.12.004
- Pastora-Bernal JM, Martín-Valero R, Barón-López FJ, Moyano NG, Estebanez-Pérez MJ. Telerehabilitation after arthroscopic subacromial decompression is effective and not inferior to standard practice: Preliminary results. *J Telemed Telecare*. 2018. doi:10.1177/1357633X17706583
- 39. Eriksson L, Lindström B, Ekenberg L. Patients' experiences of telerehabilitation at home after shoulder joint replacement. *J Telemed Telecare*. 2011. doi:10.1258/jtt.2010.100317
- 40. Pastora-Bernal JM, Martín-Valero R, Barón-López FJ. Cost analysis of telerehabilitation after arthroscopic subacromial decompression. *J Telemed Telecare*. 2018. doi:10.1177/1357633X17723367
- 41. Bain EE, Shafner L, Walling DP, et al. Use of a Novel Artificial Intelligence Platform on Mobile Devices to Assess Dosing Compliance in a Phase 2 Clinical Trial in Subjects With Schizophrenia. *JMIR mHealth uHealth*. 2017. doi:10.2196/mhealth.7030
- 42. Carnevale A, Longo UG, Schena E, et al. Wearable systems for shoulder kinematics assessment: A systematic review. *BMC Musculoskelet Disord*. 2019. doi:10.1186/s12891-019-2930-4
- 43. Wang Q, Markopoulos P, Yu B, Chen W, Timmermans A. Interactive wearable systems for upper body rehabilitation: A systematic review. *J Neuroeng Rehabil*. 2017. doi:10.1186/s12984-017-0229-y
- 44. Mejia-Hernandez K, Chang A, Eardley-Harris N, Jaarsma R, Gill TK, McLean JM. Smartphone applications for the evaluation of pathologic shoulder range of motion and shoulder scores—a comparative study. *JSES Open Access*. 2018. doi:10.1016/j.jses.2017.10.001
- 45. Chiensriwimol N, Chan JH, Mongkolnam P, Mekhora K. Monitoring frozen shoulder exercises to support clinical decision on treatment process using smartphone. In: *Procedia Computer Science*.; 2017. doi:10.1016/j.procs.2017.06.019
- 46. Viglialoro RM, Condino S, Turini G, Carbone M, Ferrari V, Gesi M. Review of the

Version: 1.4 21

- augmented reality systems for shoulder rehabilitation. *Inf.* 2019. doi:10.3390/info10050154
- 47. Carbonaro N, Lucchesi I, Lorusssi F, Tognetti A. Tele-monitoring and tele-rehabilitation of the shoulder muscular-skeletal diseases through wearable systems. In: *Proceedings of the Annual International Conference of the IEEE Engineering in Medicine and Biology Society, EMBS.*; 2018. doi:10.1109/EMBC.2018.8513371
- 48. Burns DM, Leung N, Hardisty M, Whyne CM, Henry P, McLachlin S. Shoulder physiotherapy exercise recognition: Machine learning the inertial signals from a smartwatch. *Physiol Meas*. 2018. doi:10.1088/1361-6579/aacfd9
- 49. Pan JI, Chung HW, Huang JJ. Intelligent shoulder joint home-Based self-Rehabilitation monitoring system. *Int J Smart Home*. 2013. doi:10.14257/ijsh.2013.7.5.38
- 50. Ongvisatepaiboon K, Chan JH, Vanijja V. Smartphone-based tele-rehabilitation system for frozen shoulder using a machine learning approach. In: *Proceedings 2015 IEEE Symposium Series on Computational Intelligence, SSCI 2015.*; 2015. doi:10.1109/SSCI.2015.120
- 51. Huang MC, Lee SH, Yeh SC, et al. Intelligent frozen shoulder rehabilitation. *IEEE Intell Syst.* 2014. doi:10.1109/MIS.2014.35
- 52. Correia FD, Nogueira A, Magalhães I, et al. Home-based Rehabilitation With A Novel Digital Biofeedback System versus Conventional In-person Rehabilitation after Total Knee Replacement: a feasibility study. *Sci Rep.* 2018. doi:10.1038/s41598-018-29668-0
- 53. Correia FD, Nogueira A, Magalhães I, et al. Medium-Term Outcomes of Digital Versus Conventional Home-Based Rehabilitation After Total Knee Arthroplasty: Prospective, Parallel-Group Feasibility Study. *JMIR Rehabil Assist Technol.* 2019. doi:10.2196/13111
- 54. Dias Correia F, Nogueira A, Magalhães I, et al. Digital Versus Conventional Rehabilitation After Total Hip Arthroplasty: A Single-Center, Parallel-Group Pilot Study. *JMIR Rehabil Assist Technol*. 2019;6(1):e14523. doi:10.2196/14523
- 55. Correia FD, Nogueira A, Magalhães I, et al. Home-based Rehabilitation With A Novel Digital Biofeedback System versus Conventional In-person Rehabilitation after Total Knee Replacement: a feasibility study. *Sci Rep.* 2018. doi:10.1038/s41598-018-29668-0
- 56. Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal Clinically Important Difference of the Disabilities of the Arm, Shoulder and Hand

Version: 1.4 22

Outcome Measure (DASH) and Its Shortened Version (QuickDASH). *J Orthop Sport Phys Ther*. 2014;44(1):30-39. doi:10.2519/jospt.2014.4893

Version: 1.4 23

# **ANNEX 1 - INFORMED CONSENT FORM**

Version: 1.4 24

### RESEARCH SUBJECT CONSENT FORM

Title: Digital care program for chronic shoulder tendinopathy versus

conventional physical therapy: a prospective, randomized

controlled study

Protocol No.: SH-SA-MSK-US-01

**Sponsor:** SWORD Health Technologies, Inc.

**Investigator:** Sang (Sam) Pak, PT, DPT

Assistant Professor, UCSF

Study-Related

**Phone Number(s):** 650-776-5514

**Study-Related** 

**Email Contact:** sam.pak@ucsf.edu

Ethical Approval:

### **DETAILED RESEARCH CONSENT**

You were asked for your verbal consent to take part in a research study. This document provides a concise summary of this research. It describes the key information that we believe most people need to decide whether to take part in this research. Later sections of this document will provide all relevant details.

### What should I know about this research?

Your physician explained this research to you. This form sums up that explanation.

Taking part in this research is voluntary. Whether you take part is up to you. You can choose not to take part. There will be no penalty or loss of benefits to which you are otherwise entitled.

You can agree to take part and later change your mind. There will be no penalty or loss of benefits to which you are otherwise entitled.

This research study has been thoroughly reviewed by an independent group called an Institutional Review Board ("IRB"). An IRB is a group of people who perform independent review of research studies. The protocol number given by the committee for this study is shown at the top of this information sheet.

If you don't understand, ask questions. Ask all the questions you want before you decide.

### Why is this research being done?

The purpose of this study, which is looking to enroll about 144 subjects, is to assess the clinical impact of a digital program for chronic low back pain versus conventional physical therapy.

### How long will I be in this research?

We expect that your taking part in this research will last 8 weeks. You will be asked to fill in a reassessment questionnaire once every four weeks.

### What happens to me if I agree to take part in this research?

If you decide to take part in this research study, you will be assigned at random (i.e., as if tossing a coin) to one of two groups, which we have named digital or conventional.

If you are assigned to the digital group, you will be receiving a kit with a tablet and sensors in the next few days. A mobile app on the tablet, together with the sensors, will be guiding you through exercise sessions according to a protocol specific for your condition. You will be assigned a Physical Therapist that will be monitoring your performance and progress through an online portal, and adapting the program accordingly.

You will also have access to educational texts prepared by SWORD's clinical team, which are available through a smartphone app which you have to download.

You will also have access to a cognitive behavioural therapy program. This program was designed to help you relax and give you mental tools to deal better with your condition. This program will be delivered through a weekly email, which contains a description of the objectives for the week

and a link to a pre-recorded audio session. It may also have one additional file with mental exercises to complement the sessions.

If you are assigned to the conventional group, you will be receiving two 30-minute sessions for 8 weeks, face-to-face with a Physical Therapist. These sessions will take place at the Outpatient faculty practice at UCSF. **In addition, your** assigned PT will also be communicating with you through a secure messaging system (Mychart) used at UCSF or, alternatively, through telephone check-ins (10-15 min calls, up to twice per week).

### Could being in this research hurt me?

Exercise programs can be associated with temporary pain and discomfort. If, at any point during the program, you unexpectedly experience any ill effects, contact the research team through the provided contacts: <a href="mailto:sam.pak@ucsf.edu">sam.pak@ucsf.edu</a> or 650-776-5514.

### Will it cost me money to take part in this research?

You will have access to this program at no cost to you.

### Will being in this research benefit me?

You may experience a reduction in pain, improvement in function, mood and general well-being. However, the effects vary from person to person, and we cannot promise any definite benefits to you for taking part in this research.

We cannot promise any benefits to others from your taking part in this research. However, possible benefits to others include the development of more effective evidence-based rehabilitation therapies for chronic musculoskeletal disorders.

### What other choices do I have besides taking part in this research?

Your alternative is to not take part in the research, and discuss other alternatives with your physician.

### What happens to the information collected for this research?

Your private information and your medical record will be shared with individuals and organizations that conduct or watch over this research, including:

- The research sponsor
- People who work with the research sponsor including the physical therapist
- Government agencies, such as the Food and Drug Administration
- The Institutional Review Board (IRB) that reviewed this research

We may publish the results of this research. However, we will keep your name and other identifying information confidential.

We protect your information from disclosure to others to the extent required by law. We cannot promise complete secrecy.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

Data collected in this research might be deidentified and used for future research or distributed to another investigator for future research without your consent.

### Who can answer my questions about this research?

If you have questions, concerns, or complaints, or think this research has hurt you or made you sick, talk to the research team at the phone number listed above on the first page.

### Can I be removed from this research without my approval?

The person in charge of this research can remove you from this research without your approval. Possible reasons for removal include:

- It is in your best interest
- The research is canceled by the FDA or the sponsor

We will tell you about any new information that may affect your health, welfare, or choice to stay in this research.

## What happens if I agree to be in this research, but I change my mind later?

If you decide to leave this research, contact the research team through the following contact: <a href="mailto:sam.pak@ucsf.edu">sam.pak@ucsf.edu</a> or 650-776-5514. This will not affect your access to medical care, impact your legal rights or lead to any penalty or loss of benefits to which you are otherwise entitled.

# Will I be paid for taking part in this research?

You will be paid a financial incentive of 25\$ for each electronic questionnaire you fill out and hand over to your physician.

# **Statement of Consent**

| Your signature documents your consent to take part in this research | cuments your consent to take part in this research. |
|---|---|
| Signature of adult subject capable of consent | Date |
| Signature of person obtaining consent | Date |
| Signature of testimony in case subject is unable to sign | Date |

ANNEX 2- DIGITAL THERAPEUTIC EXERCISE PROTOCOL

| Shoul | der Pain Exercise Protocol | l. Phase 1 (week 1) |
|---|---|---|
| Goals | | Precautions |
| Recovery of full range of motion (passive and active) | | |
| Decrease pain and inflammatory signs | | Do not perform loaded exercises above 70 flexion / abduction |
| Gradually increase muscular strength | | |
| | Intervention | |
| | Daily Digital Therapis | t Sessions |
| | Remote session – Assessn | nent/Deploy |
| <b>Digital Therapist Exercises</b> | Mobility | Strength 1 (External Load – RPE >8) |
| | Standing Position | )n |
| Shoulder Flexion | 2 sets of 8 reps | 2 sets of 8 reps (2/5 lbs.) (alternating) |
| Shoulder Florier | (alternating) | 2 30th 01 0 10ps (2/3 100.) (atternating) |
| Shoulder Hyperextension | 2 sets of 8 reps | |
| | (alternating) | |
| Shoulder Abduction | 2 sets of 8 reps (alternating) | 2 sets of 8 reps (5/7 lbs.) (alternating) |
| | 2 sets of 8 reps | |
| Scapular Plane Elevation | (alternating) | 2 sets of 8 reps (2/5 lbs.) (alternating) |
| Diagonal 1 Flexion | | |
| Diagonal 2 Flexion | 2 sets of 8 reps | 2 sets of 8 reps (2/5 lbs.) (alternating) |
| Diagonal 2 Picaton | (alternating) | |
| Shoulder External Rotation | 2 sets of 8 reps | 2 sets of 8 reps – Theraband (alternating |
| | (alternating) | |
| Shoulder Internal Rotation | | |
| Hand to Back | 2 sets of 8 reps | |
| | (alternating) | 2 |
| Shoulder Horizontal Abduction | | 2 sets of 8 reps (alternating) |
| Shoulder Horizontal Adduction | | |
| Shoulder External Rotation in Abduction | | 3 sets of 8 reps (5/7 lbs.) (alternating) |
|---|---|---|
| Shoulder Internal Rotation in Abduction | | |
| Scapulae Retraction with Shoulder Flexion | 2 sets of 8 reps (alternating) | |
| Scapulae Protraction with Shoulder Flexion | | |
| Arm Circles with Shoulder Flexion | | |
| Arm Circles with Shoulder Abduction | | 2 sets of 8 reps (2/5 lbs.) (alternating) |
| Chair Press-Up | | |
| Push-Up Against the Wall | | |
| Pendulum | | |
| Estimated Therapy Time | 20 min | 20 min |

| Sl | houlder Pain Exercise | e Protocol. Pha | ase 1 (weeks | 2 to 4) |
|---|---|---|---|---|
| | Goals | | | Precautions |
| Recovery of full range of motion (passive and active) Decrease pain and inflammatory signs Gradually increase muscular strength | | Do not perform loaded exercises above 70 flexion / abduction | | |
| | ] | Intervention | | |
| | | ital Therapist S<br>Remote Assess | | |
| Digital Therapist<br>Exercises | Mobility | Strength 1<br>Load – I | | Strength 2 (External Load - RPE >8) |
| | Star | nding Position | | <u> </u> |
| Forearm Supination | 2 sets of 10 reps<br>(alternating) | | | |
| Elbow Flexion | | 2 sets of (altern | - | |
| Shoulder Flexion | 2 sets of 10 reps (alternating) | 2 sets of 10<br>lbs.) (alte | • ` | |
| Shoulder Hyperextension | 2 sets of 10 reps (alternating) | | | 2 sets of 10 reps – Theraband (alternating) |
| Shoulder Abduction | 2 sets of 10 reps (alternating) | 2 sets of 10<br>lbs.) (alto | | |
| Scapular Plane Elevation | 2 sets of 10 reps (alternating) | | | 2 sets of 10 reps (2/5 lbs.) (alternating) |
| Diagonal 1 Flexion | | 2 sets of 10<br>lbs.) (alto | • ' | |
| Diagonal 2 Flexion | 2 sets of 10 reps (alternating) | | | 2 sets of 10 reps (2/5 lbs.) (alternating) |
| Shoulder External Rotation | 2 sets of 10 reps<br>(alternating) | 2 sets of<br>Theraband ( | = | |

| Cl. 11 T. 1D. | 2 sets of 10 reps | | 3 sets of 8 reps – Theraband |
|---|---|---|---|
| Shoulder Internal Rotation | (alternating) | | (alternating) |
| Hand to Back | 2 sets of 10 reps<br>(alternating) | | |
| Shoulder Horizontal | | 2 sets of 10 reps | |
| Abduction | | (alternating) | |
| Shoulder Horizontal Adduction | | | 2 sets of 10 reps (alternating) |
| Shoulder External Rotation | | 2 sets of 10 reps (5/7 | |
| in Abduction | | lbs.) (alternating) | |
| Shoulder Internal Rotation | | | 2 sets of 10 reps (5/7 lbs.) |
| in Abduction | | | (alternating) |
| Scapulae Retraction with | 2 sets of 10 reps | | |
| Shoulder Flexion | (alternating) | | |
| Arm Circles with Shoulder | | 2 sets of 10 reps (2/5 | |
| Flexion | | lbs.) (alternating) | |
| Arm Circles with Shoulder | | | 2 sets of 10 reps (2/5 lbs.) |
| Abduction | | | (alternating) |
| Chair Press-Up | | | 2 sets of 10 reps (alternating) |
| Push-Up Against the Wall | | | 2 sets of 10 reps (alternating) |
| Pendulum | | | |
| | Ly | l<br>ing Position | |
| G1 11 77 : | | 2 sets of 10 reps (2/5 | |
| Shoulder Flexion | | lbs.) (alternating) | |
| Chauldon Fretzers I. D. 444 | | | 2 sets of 10 reps (2/5 lbs.) |
| Shoulder External Rotation | | | (alternating) |
| Shoulder Internal Rotation | | 2 sets of 10 reps (2/5 | |
| Shoulder internal Rotation | | lbs.) (alternating) | |
| <b>Estimated Training Time</b> | 29 min | 29 min | 28 min |

| Shoulder Pain Exercise Protocol. Phase 2 (Weeks 5 to 8) | | | | |
|---|---|---|---|---|
| Goals | | | Precautions | |
| Range of motion conservation | Range of motion conservation | | | |
| Global muscular strengthening | g in | | | |
| asymptomatic range of movement, | focusing | Do no | ot perform push-ups on the f | loor in case of complete |
| on: | | Do no | rotator cuff tears (use in | _ |
| - Rotator cuff | | | ` | , |
| - Scapular stabilizers | | | | |
| - Deltoids | | | | |
| | | Interven | ntion | |
| | Daily I | Digital Ther | apist Sessions | |
| | 8 W | eek Remote | Assessment | |
| Digital Thomasist Evansises | Мо | h:1:4 | Strength 1 (External | Strength 2 (External |
| Digital Therapist Exercises | IVIO | bility | Load – RPE >8) | Load – RPE >8) |
| | | Standing P | Position | |
| Shoulder Flexion | 2 sets c | of 10 reps | 2 sets of 10 reps (5/7 | |
| Shoulder Flexion | (alter | nating) | lbs.) (alternating) | |
| | | | | 2 sets of 10 reps |
| Shoulder Hyperextension | | | | (Theraband) |
| | | | | (alternating) |
| Shoulder Abduction | 2 sets c | of 10 reps | 2 sets of 10 reps (5/7 | |
| Shoulder Abduction | (alter | rnating) | lbs.) (alternating) | |
| Scapular Plane Elevation | 2 sets c | of 10 reps | | 2 sets of 10 reps (5/7 |
| Scapulal Flane Elevation | (alternating) | | | lbs.) (alternating) |
| Diagonal 1 Flexion | 2 sets c | of 10 reps | 2 sets of 10 reps (5/7 | |
| Diagonal I Fiexion | (alter | rnating) | lbs.) (alternating) | |
| Diagonal 2 Flevion | 2 sets c | of 10 reps | | 2 sets of 10 reps (5/7 |
| Diagonal 2 I tonion | Diagonal 2 Flexion (alterna | | | lbs.) (alternating) |

| Shoulder External Rotation | 2 sets of 10 reps<br>(alternating) | 2 sets of 10 reps (Theraband) (alternating) | |
|---|---|---|---|
| Shoulder Internal Rotation | | | 2 sets of 10 reps (Theraband) (alternating) |
| Hand to Back | 2 sets of 10 reps<br>(alternating) | | |
| Shoulder Horizontal Abduction | | 2 sets of 10 reps (Theraband) (alternating) | |
| Shoulder Horizontal Adduction | | | 2 sets of 10 reps (Theraband) (alternating) |
| Shoulder External Rotation in | 2 sets of 10 reps | 2 sets of 10 reps (5/7 | |
| Abduction | (alternating) | lbs.) (alternating) | |
| Shoulder Internal Rotation in | 2 sets of 10 reps | | |
| Abduction | (alternating) | | |
| Scapulae Retraction with | 2 sets of 10 reps | | |
| Shoulder Flexion | (alternating) | | |
| Scapulae Protraction with Shoulder Flexion | | | |
| Arm Circles with Shoulder | | 2 sets of 10 reps (5/7 | |
| Flexion | | lbs.) (alternating) | |
| Arm Circles with Shoulder Abduction | | | 2 sets of 10 reps (5/7 lbs.) (alternating) |
| Chair Press-Up | | | 2 sets of 10 reps<br>(consecutive) |
| Push-Up Against the Wall | | | 2 sets of 10 reps (alternating) |
| Pendulum | | | |

| Lying Position | | | |
|---|---|---|---|
| Shoulder Flexion | | 2 sets of 10 reps (5/7 | |
| | | lbs.) (alternating) | |
| Shoulder Abduction | | 2 sets of 10 reps (5/7 | |
| | | lbs.) (alternating) | |
| Shoulder External Rotation | | | |
| Shoulder Internal Rotation | | | |
| Shoulder Horizontal Abduction | | | 2 sets of 10 reps (5/7 |
| | | | lbs.) (alternating) |
| Arm Circle with Shoulder | | 2 sets of 10 reps (5/7 | |
| Flexion | | lbs.) (alternating) | |
| Arm Circle with Shoulder | | | 2 sets of 10 reps (5/7 |
| Abduction | | | lbs.) (alternating) |
| Estimated Training Time | 29 min | 29 min | 27 min |

ANNEX 3- CONVENTIONAL PT INTERVENTION PROTOCOL

The co-investigators are encouraged to use the McClure's staged based rehabilitation therapy (STAR) classification (see Table 1) as a *guide* but not necessarily as a prescriptive manner to select interventions. Instead, the co-investigators will reference their use interventions categorized based on commonly practiced in an outpatient physical therapy setting (see Table 2).

McClure's stage-based rehabilitation therapy (STAR) intervention approach is based on the Irritability of the patient's condition. Assessments of symptoms of Irritability are gathered from the patient's history and findings from the examination. Table 1 represents a guided approach to STAR for the chronic shoulder pain population and the type of interventions used. Table 2 describes the type of commonly used physical therapy interventions that could be used in the cohorts.

## Guideline to help determine the stage of Irritability is based on both history and examination findings\*

| High | Moderate | Low |
|---|---|---|
| • Pain >= 7/10 | • Pain (4-6/10) | • Pain (<= 3/10) |
| • Consistent night or | Intermittent night or rest pain | Absent night or rest pain |
| resting pain | Pain at end of range | Minimal pain with overhead |
| • Pain before end of range | AROM and PROM close | • AROM = PROM |
| • AROM < PROM | Moderate disability | Low disability |
| High disability | | |
| Approach: Minimize | Approach: Mild-moderate physical | Approach: Mod-high physical |
| physical stress | stress | stress |
| • Activity | Basic-level functional | High-demand functional |
| modification | activity restoration | activities |

<sup>\*</sup>Taken from Staged approach (STAR) for rehabilitation classification by McClure et al.

Table 1. McClure's staged approach to shoulder intervention based on different impairments

| Impairments | Irritability | Intervention | Examples of |
|---|---|---|---|
| | | Approaches | Intervention** |
| Restricted passive mobility | Low | • ROM | Aggressive active and |
| due to joint/muscle/neural | | Stretching | passive stretches (e.g., |
| tissues | | • manual therapy: | sleeper stretches; |
| | | tolerable stretch | foam roller T's, Y's, |
| | | sensation at end- | I's; Doorway stretch) |
| | | range | |
| | | Hold longer | |
| | | duration and | |
| | | frequency | |
| Restricted passive mobility | Moderate | • ROM | Active and passive |
| due to joint/muscle/neural | | Stretching | stretches (e.g., gentle |
| tissues | | Comfortable end- | sleeper stretches; |
| | | range manual | Foam roller T's, Y's, |
| | | therapy | I's; modified to ½ to |
| | | | full foam roller T's, |
| | | | Y's, I's; Modified |
| | | | doorway stretch) |
| Restricted passive mobility | High | • ROM | AAROM/PROM |
| due to joint/muscle/neural | | Stretching | (e.g., ½ roller; towel |
| tissues | | Pain-free manual | rolls; wall crawl) |
| | | therapy | |
| | | Avoid end-range | |
| Excessive passive mobility | High | Protect joint/tissue | Gentle isometrics |
| | | from end-range | |

| Impairments | Irritability | Intervention | Examples of |
|---|---|---|---|
| | | Approaches | Intervention** |
| | | Manual therapy to | Parascapular |
| | | reduce pain | strengthening |
| Excessive passive mobility | Mod | Develop active control in mid-range while avoiding end- range in basic activity Address | Isometrics to isokinetic (e.g., ER/IR/ABD/Flex, parascapular stabs) |
| | | hypomobility of adjacent joints or tissues | |
| Excessive passive mobility | Low | Develop active control during full- range, high-level functional activity Address hypomobility of adjacent joints or tissues | Isokinetic to dynamic (e.g., ER/IR/ABD/Flex, parascapular stabs) |
| Neuromuscular weakness<br>due to atrophy, disuse,<br>and/or deconditioning | High | AROM within pain-<br>free ranges | <ul> <li>AAROM/AROMS via Pulleys, table slides </li> <li>Isometrics (e.g. ER/IR/ABD/Flex, parascapular stabs) </li> </ul> |

| Impairments | Irritability | Intervention | Examples of |
|---|---|---|---|
| | | Approaches | Intervention** |
| Neuromuscular weakness due to atrophy, disuse, and/or deconditioning | Mod | Light or moderate resistance to fatigue Mid-ranges | <ul> <li>Isometrics to isokinetic</li> <li>Rotator cuff strengthening (ER/IR) in neutral to variations of ABD via weights or T-band (i.e., ER/IR/ABD/Flex, parascapular stabs)</li> </ul> |
| Neuromuscular weakness due to atrophy, disuse, and/or deconditioning | Low | Moderate or high resistance to fatigue Include end-ranges | <ul> <li>Isokinetic to dynamic resistive movements</li> <li>Rotator cuff strengthening (ER/IR/Flex/ABD) in progression from neutral to variations of movements via weights or T-band</li> </ul> |
| Neuromuscular weakness associated with poor motor control or neural activation | High | <ul> <li>AROM within painfree ranges</li> <li>Biofeedback,</li> <li>Neuromuscular electrical stimulation, or other activation strategies</li> </ul> | <ul> <li>Isometrics (e.g.,<br/>ER/IR, parascapular<br/>stabs)</li> <li>Mirror/manual cue<br/>feedback for<br/>AROM/AAROM;<br/>Scapular<br/>clock exercises</li> </ul> |

| Impairments | Irritability | Intervention | Examples of |
|---|---|---|---|
| | | Approaches | Intervention** |
| Neuromuscular weakness | Mod | Basic movement | • Isometrics to |
| associated with poor motor | | training with | isokinetic (e.g., |
| control or neural | | emphasis on | ER/IR, parascapular |
| activation | | quality/precision | stabs) |
| | | rather than | loaded motor control |
| | | resistance according | exercises with mirror |
| | | to motor learning | feedback |
| | | principles | |
| Neuromuscular weakness | Low | High-demand | Isokinetic to |
| associated with poor motor | | movement training | dynamics (e.g., |
| control or neural | | with emphasis on | ER/IR, parascapular |
| activation | | quality rather than | stabs) |
| | | resistance according | • Progressive loaded |
| | | to motor learning | motor control |
| | | principles | exercises with mirror |
| | | | feedback |
| Restricted tolerance to | High | Maximum joint or | Patient education |
| functional activity | | tissue protection | (e.g., anatomy; |
| | | from end-range | biomechanics; |
| | | Advocate use of | supplemental |
| | | unaffected regions | youtube videos; |
| | | | Tissue healing |
| | | | timelines; Pain |
| | | | science) |
| | | | • CBT |
| | | | Graded activity and |
| | | | graded exposure |

| Impairments | Irritability | Intervention | Examples of |
|---|---|---|---|
| | | Approaches | Intervention** |
| | | | exercises / functional activities |
| Restricted tolerance to functional activity | Mod | Progressively engage in basic functional activity | <ul> <li>Patient education (e.g., anatomy; biomechanics; supplemental youtube videos; Tissue healing timelines; Pain science)</li> <li>CBT</li> <li>Progress graded activity and graded exposure exercises / functional activities</li> </ul> |
| Restricted tolerance to functional activity | Low | Progressively engage in basic functional activity | <ul> <li>Patient education <ul> <li>(e.g., anatomy;</li> <li>biomechanics;</li> <li>supplemental</li> <li>youtube videos;</li> <li>Tissue healing</li> <li>timelines; Pain</li> <li>science)</li> </ul> </li> <li>CBT</li> <li>Progress graded <ul> <li>activity and graded</li> </ul> </li> </ul> |

| Impairments | Irritability | Intervention | Examples of |
|---|---|---|---|
| | | Approaches | Intervention** |
| | | | exposure exercises / |
| | | | functional activities |
| Limited patient | Low/Mod/High | Select appropriate | Patient education |
| understanding of condition | | patient education | (e.g., anatomy; |
| leading to inappropriate or | | | biomechanics; |
| avoidance of activity | | | supplemental |
| | | | youtube videos; |
| | | | Tissue healing |
| | | | timelines; Pain |
| | | | science) |
| | | | • CBT |
| | | | Motivational |
| | | | interviews |

<sup>\*\*</sup>Not a comprehensive list of interventions/exercises

**Table 2. General Category of Physical Therapy Interventions** 

| Intervention | Description | Type of Interventions | Examples of |
|---|---|---|---|
| Categories | | | Intervention** |
| Therapeutic | Systematically planned | Flexibility | • Strengthening - ER/IR |
| Exercises | performance of bodily movement, postures, | <ul><li>Strengthening</li><li>Endurance</li></ul> | in neutral position with T-band |
| | physical activities relevant to patient's condition* | <ul> <li>Neuromuscular reeducation</li> <li>Functional task training</li> </ul> | <ul> <li>Flexibility - Wall slides in standing</li> <li>Functional activities training</li> </ul> |
| Patient Education | Informing, educating, training patients related to their condition | <ul> <li>Disease condition</li> <li>Anatomy</li> <li>Activity modification</li> <li>Ergonomics</li> <li>Cognitive Behavior Therapy/Motivational Interview</li> <li>Symptom management</li> </ul> | <ul> <li>Patient education on glenohumeral joint and surrounding tissues</li> <li>Precautions of activities for shoulder joint</li> </ul> |
| Manual Therapy | Skilled passive movements of joints/soft tissue | <ul> <li>Joint mobilization</li> <li>Soft tissue mobilization</li> <li>Neural tissue mobilization</li> <li>Therapeutic massage</li> </ul> | <ul> <li>Passive accessory motion of anterior- posterior of glenohumeral joint</li> <li>Passive physiological motion of glenohumeral joint</li> </ul> |

| | | | Myofascial |
|---|---|---|---|
| | | | decompression |
| | | | (Cupping) |
| Biophysical | Use of a broad group | Electric Stimulation | Electrical muscle |
| Agents/Modalities | of modalities for | Ultrasound | stimulation (EMS) |
| | therapeutic purposes | Heat/Ice | Neuromuscular |
| | | Taping | electrical stimulation |
| | | Biofeedback | (NMES) |

<sup>\*</sup>Definition is taken from APTA Guide to Physical Therapists Practice

<sup>\*\*</sup>Not a comprehensive list of interventions/exercises